CLINICAL TRIAL: NCT01747993
Title: Tamsulosin to Facilitate Early Catheter Removal After Urinary Retention in Older Women Hospitalized for an Acute Medical Condition
Brief Title: Tamsulosin for Urinary Retention in Hospitalized Older Women
Acronym: TAMSU
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P 101005; AOR11001 (Other: Assistance Publique)
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-10

CONDITIONS: Urinary Retention
Keywords: Urinary retention; urinary catheterization; alpha blocking agents; women; elder
MeSH Terms: conditions — Urinary Retention | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tamsulosin (Experimental): Tamsulosin (0.4 mg/j) (1 tablet / day for 6 days)
  Interventions: Drug: Tamsulosin (0.4 mg/j)
- placebo (Placebo Comparator): 1 tablet / day for 6 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin (0.4 mg/j) — (1 tablet / day for 6 days)
  Arms: tamsulosin
Drug: Placebo — (1 tablet / day for 6 days)
  Arms: placebo

SUMMARY:
Catheter-associated urinary infections are the most common hospital-acquired infections and can be prevented by early catheter removal. This study evaluates tamsulosin to reduce the failure of early catheter removal has been studied in elderly women hospitalized for an acute condition and experiencing acute urinary retention: 448 women 75-year old or more without an anatomical or neurological cause of urinary retention will be randomized to a 6 days course of tamsulosin 0.4 mg or placebo. Catheter removal will be attempted after the third dose of tamsulosin and the need to replace another catheter within 72 hours will define a failed attempt.

DETAILED DESCRIPTION:
Background: Urinary tract infections are the most frequent hospital-acquired infections. A majority is catheter-associated and the main risk factor is the duration of catheterization. Early removal is therefore a priority. Treatment with alpha-blockers in men with acute urinary retention due to prostatic disease increases the rate of successful early catheter removal. No intervention has been studied in elderly women in whom urinary retention is usually favored by an acute health issue. However, alpha-blockers have proved effective in other circumstances, as the prevention of acute urinary retention after hysterectomy and the treatment of chronic voiding disorders.

Objective: To evaluate the benefit of tamsulosin for 6 days in older women hospitalized for an acute medical condition and experiencing urinary retention.

Primary endpoint: Rate of failed early catheter removal (day 3), requiring placement of another catheter within the following 72 hours.

Secondary endpoints: rate of hospital-acquired urinary tract infections, rate of hypotension, length of hospitalization.

Design: Double-blind and multicentric randomized controlled trial (tamsulosin 0.4 mg/day or placebo orally for 6 days).

Number of patients: We assume a 40% failure rate of early catheter removal in the placebo group. Expecting a 10% dropout rate, 448 patients need to be randomized to show a reduction of this rate by one third in the tamsulosin group with two-sided alpha level at 5% and beta level at 20%.

Inclusion criteria: 75-year or older women hospitalized in an internal medicine or geriatric ward and with a bladder catheter for less than 48 hours for acute urinary retention.

Non-inclusion criteria: chronic urinary retention; acute retention with an anatomical (pelvic tumor, pelvic surgery) or neurological cause (peripheral neuropathy, spinal cord compression, multiple sclerosis, amyotrophic lateral sclerosis, Parkinson's disease); catheter placed for another indication (pressure ulcer protection, urine output monitoring); patients at the end of life; contra-indication to alpha-blockers.

Course of the study: The patient receives a treatment dose in the evening inclusion (day 0) and the five following evenings. The catheter is removed after the third dose, between midnight and noon. The patient is followed up until day 12.

Total time: 36 months (35 months of inclusion + 12 days of participation per patient).

Number of participating centers: 8 Expected number of inclusions per month and center: 2-4

ELIGIBILITY:
Inclusion Criteria:

* 75-year or older women hospitalized in an internal medicine or geriatric ward and with a bladder catheter for less than 48 hours for acute urinary retention.

Exclusion Criteria:

* chronic urinary retention;
* acute retention with an anatomical (pelvic tumor, pelvic surgery) or neurological cause (peripheral neuropathy, spinal cord compression, multiple sclerosis, amyotrophic lateral sclerosis, Parkinson's disease);
* catheter placed for another indication (pressure ulcer protection, urine output monitoring);
* patient at the end of life;
* contra-indication to alpha-blockers.

Min Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
early catheter removal failure | between days 3 and 6
  need to replace a catheter within 72h following day 3 catheter removal

SECONDARY OUTCOMES:
hospital-acquired urinary tract infection | between days 1 and 12
  any symptomatic urinary tract infection proved by urine culture
orthostatic hypotension | days 1 to 6
  blood pressure drop > 20/10 mmHg between lying and standing
length of hospitalization | from day 1
  number of days in the ward where the patient was enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bouvard, MD, Principal Investigator — Assistance Publique
Locations (1):
- Service de médecine interne, Hôpital Tenon, Paris, France